CLINICAL TRIAL: NCT02243813
Title: Effects of Psilocybin-facilitated Experience on the Psychology and Effectiveness of Professional Leaders in Religion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00036973
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Psilocybin; Pharmacologic Actions; Psychotropic Drugs
MeSH Terms: interventions — Psilocybin

ARMS (2):
- Delayed Participation (Experimental): Participants will begin the psilocybin intervention 6 months after study enrollment.
  Interventions: Drug: Psilocybin
- Immediate Participation (Experimental): Participants will begin psilocybin intervention immediately after study enrollment.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive 20 mg/70 kg of psilocybin in the first session and will receive either 20 or 30 mg/70 kg in the second session.

SUMMARY:
The current protocol is a pilot study of the effects and possible utility of psilocybin-facilitated experiences for professional religious leaders.

ELIGIBILITY:
Inclusion criteria:

* Have given written informed consent
* College graduation or equivalent and graduate/professional training.
* Recognized leadership position in a well-established religious organization; professional activities must include significant time interacting with those seeking religious/spiritual guidance or support.
* Be healthy and psychologically stable as determined by screening for medical and psychiatric problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* During the next year there is no foreseen likelihood for a major potentially life-altering event for her or himself or a close family member (e.g. retirement or major career change for the volunteer; life-threatening illness of a spouse or child of the volunteer)
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of psilocybin session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, 24 hours before and after each drug administration. The exception is caffeine. Participants will be required to be either a non-smoker or a non-daily smoker.
* Agree not to take any Pro-re-nata (PRN) medications on the mornings of drug sessions
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.

General medical exclusion criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant Electrocardiogram (ECG) abnormality (e.g., symptomatic atrial fibrillation), or Transient Ischemic Attack (TIA) in the past year
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting pharmacological effect on serotonin neurons or medications that are Mono amine Oxidase (MAO) inhibitors. For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* More than 20% outside the upper or lower range of ideal body weight according to Metropolitan Life height and weight table

Psychiatric Exclusion Criteria:

* Current or past history of meeting Diagnostic and Statistics Manual (DSM)-5 criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder
* Current or past history within the last 5 years of meeting DSM-5 criteria for alcohol or substance use disorder (excluding caffeine and nicotine) or severe major depression
* Have a first or second-degree relative with Schizophrenia, Psychotic Disorder (unless substance induced or due to a medical condition), or Bipolar I or II Disorder
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Interim Questionnaire | 6 months after enrollment
  This questionnaire asks about experiences and changes in attitudes, mood and behavior that occurred during the past 5 months. The questionnaire includes questions about salient spiritual experiences, changes in spiritual practices, changes in attitudes, moods, social interactions, and other behaviors related to participants' religious/spiritual vocation.

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, Ph.D., Principal Investigator — JHUSOM
Locations (1):
- Behavioral Biology Research Center, Johns Hopkins Bayview, Baltimore, Maryland, United States

REFERENCES:
- See also: Study Flyer — http://www.religiousleaderstudy.org